CLINICAL TRIAL: NCT02768233
Title: Medication-overuse Headache: The Effect of a Patient Educational Programme as an add-on to Standard Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Louise Schlosser Mose, PhD student, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20140114
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Secondary Headache Disorders; Medication-overuse Headache
Keywords: Medication-overuse Headache; Educational Programme; Personality Profiles
MeSH Terms: conditions — Headache Disorders, Secondary

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational programme (Experimental): Group 1: Educational programme + standard treatment
  Interventions: Behavioral: Educational programme
- Standard treatment (No Intervention): Standard treatment

INTERVENTIONS:
Behavioral: Educational programme — The 6-session educational programme is based on theory of motivational interviewing, and patients can choose between individualized education or education in groups. The standard treatment consists of withdrawal and consultations by neurologist.
  Arms: Educational programme

SUMMARY:
The aim of this study is to evaluate the influence of personality profiles in patients with MOH and to evaluate the effect of a custom-made educational programme as an add-on to standard treatment as compared to standard treatment alone in MOH patients using a randomized controlled trial (RCT) design.

DETAILED DESCRIPTION:
Worldwide, two percent of the population suffers from medication-overuse headache (MOH), a paradox condition where the headache is caused by overuse of headache medication. Common treatment is withdrawal, but there is no consensus on what constitutes the best treatment.

The study consists of a RCT with MOH patients randomized to standard treatment versus standard treatment + a 12-week, 6-session educational programme as add-on. The programme is based on theory of motivational interviewing, and patients can choose between individualized education or education in groups.

Primary endpoint: Headache frequency measured by self-reported headache diary on number of days with headache pre-vious month. Secondary endpoints: NEO-FFI-3 personality test, coping strategies, pain intensity, bothersomeness, patient satis-faction and reported medication intake.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with medication-overuse headache (MOH) by neurologist (The International Classification of headache Disorders).
* Completed withdrawal (hospitalized of 8 days or at home).
* Age 18-65 years
* Understand and speak Danish

Exclusion Criteria:

* Comorbidity (e.g. whiplash, rheumatism which needs analgesic treatment
* Mental health disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Headache frequency measured by self-reported headache diary on number of days with headache previous month | baseline-36 weeks follow-up

SECONDARY OUTCOMES:
NEO-FFI-3 personality test | Baseline
  self reported. 63 items. Each item scores using a 5 point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree)
Coping Strategies | Baseline, Post intervention (16 weeks), Follow-up (36 weeks)
  CSQ Questionnaire (Scale ranging from 0 (never) to 6 (always)
Pain Intensity | Baseline, Post intervention (16 weeks), Follow-up (36 weeks)
  VAS (0: No pain, 10: Pain as bad as it can be)
Bothersomeness | Baseline, Post intervention (16 weeks), Follow-up (36 weeks)
  VAS (0: No bothersomeness, 10: Bothersomeness as bad as it can be)
Patient satisfaction | Baseline, Post intervention (16 weeks), Follow-up (36 weeks)
  Questionnarire
Medication intake | baseline, Post intervention (16 weeks) and Follow-up (36 weeks)
  self reported intake (type, name of medication, dosis)

CONTACTS AND LOCATIONS:
Overall Officials: Louise S. Mose, MHS, Principal Investigator — Hospital of South West Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mose LS, Pedersen SS, Jensen RH, Gram B. Medication-overuse headache: The effect of a patient educational programme-A randomized controlled trial. Eur J Pain. 2020 Feb;24(2):435-447. doi: 10.1002/ejp.1500. Epub 2019 Nov 21. PMID 31661579